CLINICAL TRIAL: NCT01295892
Title: Chronic Effects of Estrogen in Microcirculation and Insulin Resistance in Postmenopausal Obese Women
Brief Title: Chronic Effects of Estrogen in Microcirculation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Luiz Guilherme Kraemer de Aguiar, Chronic Effects of Estrogen in Microcirculation and Insulin Resistance in Postmenopausal Obese Women, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: pkvw6k
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Postmenopausal Symptoms
Keywords: menopause; obesity; capillary; microcirculation; estrogen; Microvascular Function
MeSH Terms: conditions — Obesity | interventions — Estrogens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo (transdermal gel)
  Interventions: Drug: Estrogen
- Estrogen (Experimental): 1mg of 17B-estradiol/day (transdermal gel)
  Interventions: Drug: Estrogen

INTERVENTIONS:
Drug: Estrogen — transdermal 17-β-estradiol 1mg/day during three months

SUMMARY:
This study aims to evaluate the chronic effects of estrogen on microcirculation, inflammatory biomarkers, hormonal status, plasma viscosity and biochemical tests in postmenopausal obese women after three months of follow-up intervention.

DETAILED DESCRIPTION:
Estrogens exert pleiotropic actions on the cardiovascular system through binding to estrogen receptors. Traditionally, estrogen receptors have been recognized as transcription factors regulating the expression of target genes, however, numerous studies have revealed rapid actions of estrogen in different systems, so-called 'extranuclear actions'. At this level, estrogen triggers rapid vasodilatation, exerts anti-inflammatory effects, regulates vascular cell growth and migration, and confers protection to cardiomyocytes. Our aims are to investigate estrogen´s chronic effects on microcirculation.

The study will assess the potential benefits of estrogens on: chronic low-grade inflammation, metabolic profile, microcirculation and blood rheology. Postmenopausal obese women will be randomly submitted to estrogen (transdermal 17-β-estradiol 1mg/day) or placebo therapy during three months in a double-blind fashion. At baseline and after intervention, nailfold videocapillaroscopy, laser-Doppler flowmetry and venous occlusion plethysmography, inflammatory biomarkers, hormonal status, metabolic profile, plasma viscosity and anthropometrical measures will be assessed in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* History of natural menopause defined by the absence of menses for at least 12 months and a serum concentration of FSH > 35 IU/L
* BMI between 27 to 34.9 kg/m²
* Non-smokers
* Not on use of any hormones or supplements for a minimum of 6 months prior to the study
* No absolute contraindications to the use of physiological replacement doses of estrogen

Exclusion Criteria:

* Renal disease, coronary or peripheral vascular diseases, haematologic or hepatic diseases
* Diabetes mellitus, glucose intolerance or altered fasting glucose

Ages: 48 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
functional capillary density by videocapillaroscopy(number of perfused capillaries on the studied skin area) | 03 months

SECONDARY OUTCOMES:
blood viscosity(the values are expressed in centipoises) | 03 months
  evaluate the change in blood viscosity after 3 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Diogo Panazzolo, Principal Investigator — Rio de Janeiro State University
Locations (1):
- Laboratorio de Pesquisas Clinicas e Experimentais em Biologia Vascular, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] da Silva LH, Panazzolo DG, Marques MF, Souza MG, Paredes BD, Nogueira Neto JF, Leao LM, Morandi V, Bouskela E, Kraemer-Aguiar LG. Low-dose estradiol and endothelial and inflammatory biomarkers in menopausal overweight/obese women. Climacteric. 2016 Aug;19(4):337-43. doi: 10.1080/13697137.2016.1180676. Epub 2016 May 12. PMID 27170466